CLINICAL TRIAL: NCT02444299
Title: An Observational Cohort Study Evaluating the Safety and Performance of Aequalis Resurfacing Head Implant in a Consecutive Series of Patients With Shoulder Arthroplasty
Brief Title: Aequalis Resurfacing Head Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 0908-T-RESURF-RM
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2018-04

CONDITIONS: Localized, Primary Osteoarthritis; Post-traumatic Arthrosis of Other Joints, Shoulder Region; Avascular Necrosis of the Head of Humerus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Shoulder hemi-arthroplasty

SUMMARY:
Aequalis® Resurfacing Head implant is a range of shoulder arthroplasty device available for the treatment of various shoulder pathologies. It received CE Mark in June 2007.

The aim of this study is to collect immediate medium and long term data on performance and safety of the implant, retrospectively as well as prospectively, from a consecutive series of patients to assess the patients' outcomes and functional status.

DETAILED DESCRIPTION:
Resurfacing head implants allow restoring of the normal joint mechanics and stability of the shoulder with minimal bone resection and low peripheral fracture risk, while preserving humeral bone stock. Non cemented head implants also allow for an easy re-intervention if needed. The success of resurfacing implants largely depends on the etiology, with the best results in primary shoulder arthrosis, and the worst in post-traumatic and cuff-tear arthropathy.

The Aequalis® Resurfacing Humeral Head is designed to restore the humeral head. It shares the same indications as shoulder arthroplasty in general, including the various types of arthritis and conditions resulting in loss of joint cartilage, joint incongruity, pain, and stiffness. Resurfacing humeral head implants allow minimal bone resection while preserving humeral bone stock as compared to standard anatomic humeral implants.

However, few data are available on mid-term effects of the resurfacing head implant developed by Tornier. This Post-Marketing study is implemented for the Aequalis® Resurfacing Head in shoulder arthroplasty to collect medium and long-term clinical data on performance and safety. It is designed to collect data from consecutive series in European patients for at least 12 months of follow-up and up to 10 years. If possible, the study duration and collection of information will be prolonged. Further follow-up can be implemented, by amendments.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received an Aequalis® Resurfacing Head implant as per the manufacturer's instructions (including the recommended indication): degenerative indication such as primary osteoarthritis, secondary osteoarthritis (post-traumatic post instability), avascular osteonecrosis of the humeral head ;
* with a functional rotator cuff ;
* has clinical and radiographic follow-up data available ;
* is informed about the study and has provided Informed Consent as applicable.

Exclusion Criteria:

* Patient with proximal humeral fracture,
* previous history of infection,
* rotator cuff tear, cuff tear arthropathy,
* significant bone loss of the glenoid (more than 25% of the articular surface),
* nerve palsy,
* revision arthroplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from 6 centers in Europe where shoulder arthroplasty with Aequalis® Resurfacing Head is performed.
  The first 100 patients treated in the centers will be included then followed-up, until the 10 years follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | up to 10-year follow-up
  Number or device or procedure related adverse events

SECONDARY OUTCOMES:
Change from baseline and previous visit in Constant Murley score | at 3-month, 1, 2, 5, 10 years follow-up
Change from baseline and previous visit in Range Of Motion | at 3-month, 1, 2, 5, 10 years follow-up
  Passive and active Abduction, external rotation and internal rotation will be assessed.
Change from baseline and previous visit in SSV. | at 3-month, 1, 2, 5, 10 years follow-up
  The Subjective Shoulder Value (SSV) is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.

OTHER OUTCOMES:
Timely evaluation of fixation and migration of the implant. | at 3-month, 1, 2, 5, 10 years follow-up
  Presence of radiolucent line(s) around the implant (Radiological imaging : X-Rays of MRI).
Timely evaluation of glenoid status. | at 3-month, 1, 2, 5, 10 years follow-up
  Radiological imaging (X-Rays or MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Lionel NEYTON, MD, Principal Investigator — Centre Orthopédique Santy, Lyon, FR